CLINICAL TRIAL: NCT03429660
Title: French Adult Primary Immune Thrombocytopenia: a pHarmacoepidemiological Study
Brief Title: French Adult Primary Immune Thrombocytopenia
Acronym: FAITH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31-14-7439B
Record Dates: First submitted 2017-02-21; First posted 2018-02-12 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Thrombocytopenia
Keywords: Disease epidemiology; Risk assessment; Drug utilisation study; Effectiveness evaluation
MeSH Terms: conditions — Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Data to be collected are :
  - Medical information on Immune Thrombocytopenia treatment
  Interventions: Other: Medical information

INTERVENTIONS:
Other: Medical information — The information collected are about :
  * Introduction or non-introduction of treatment
  * Cumulative dose of treatment
  * Drug dispensation and withdrawal
  * Hospitalization reason
  * Safety information
  * Demographic data (date of death)

SUMMARY:
Primary immune thrombocytopenia (ITP) is rare. First-line treatment is corticotherapy. Then, several second-line treatments (SLT) are available: splenectomy, off-label rituximab and thrombopoietin-receptor agonists since 2009. The compared efficacy and safety on clinical events in the long-term are unknown. The main objective of the FAITH study is to build the cohort of all treated adult persistent (≥3 months) primary ITP patients in France, to assess the benefit-to-risk ratio of SLT in real-life practice. Data source is the database of French Health Insurance System (SNIIRAM) which covers the entire French population. It collects demographic, chronic disease, hospitalization and drug dispensing data. All patients with ITP were extracted from 2009 to 2012, and then every year for 10 years. The investigator will build the cohort from raw data. Outcomes (death, hospitalization, drug dispensing) will be compared according to SLT, with controls from the general population and untreated patients.

ELIGIBILITY:
Inclusion Criteria:

* Incident case of immune thrombocytopenia or control patient

Exclusion Criteria:

* Patient not registered in the database between 2009 and 2012

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of patient registred in national administrative french database
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-10; Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Exposition or non exposition to available immune thrombocytopenia persistent | up to 10 years
  Data will be extracted until the end of study

SECONDARY OUTCOMES:
Mortality as assessed date of death collected in the database | Each year until 10 years
  Data will be extracted every year of the study until the end of study
Number of hospitalization for bleeding in the database | Each year until 10 years
  Number of hospitalization for bleeding will be extract from database every year
Safety of treatment for infections | Each year until 10 years
  Number of infections is represented by number of hospitalization and antibiotics dispensation and will be extract from database every year
Safety of treatment for cardio-vascular events | Each year until 10 years
  Number of hospitalization for cardio-vascular events will be extract from database every year
Safety of treatment for thrombo-embolic events | Each year until 10 years
  Number of hospitalization for thrombo-embolic events will be extract from database every year

CONTACTS AND LOCATIONS:
Overall Officials: Maryse LAPEYRE-MESTRE, PHD, Study Director — University Hospital of Toulouse
Locations (1):
- University Hospital of Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided